CLINICAL TRIAL: NCT02635867
Title: Clinical Comparison of Vital Pulp Capping Restorative Protocols: A Randomized Controlled Double-Blind, Prospective Study
Brief Title: Clinical Comparison of Vital Pulp Capping Restorative Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Ana Bedran-Russo, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2014-1163
Record Dates: First submitted 2015-12-08; First posted 2015-12-21 (Estimated); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2022-12

CONDITIONS: Deep Dental Caries
Keywords: vital pulp; reversible pulpitis; pulp capping; deep cavity; Management of Deep Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (5):
- Indirect pulp capping therapy-Resin-modified calcium silicate - TheraCal (Active Comparator): Resin modified calcium silicate-TheraCal (light curable)
  Interventions: Procedure: Indirect Pulp capping-Resin-modified calcium silicate - TheraCal
- Indirect pulp capping therapy- - Calcium hydroxide - Dycal (Active Comparator): Calcium hydroxide - Dycal
  Interventions: Procedure: Indirect Pulp capping-Calcium hydroxide - Dycal
- Indirect pulp capping therapy-- Resin-based dentin bonding agent (Active Comparator): Resin-based dentin bonding agent-Self etching adhesive
  Interventions: Procedure: Indirect Pulp capping-Resin-based dentin bonding agent
- Direct pulp capping therapy-Resin-modified calcium silicate - TheraCal (Active Comparator): Resin modified calcium silicate-TheraCal (Light curable)
  Interventions: Procedure: Direct Pulp capping-Resin-modified calcium silicate - TheraCal
- Direct pulp capping therapy-Resin-modified calcium silicate - Calcium hydroxide - Dycal (Active Comparator): - Calcium hydroxide - Dycal
  Interventions: Procedure: Direct Pulp capping-Calcium hydroxide - Dycal

INTERVENTIONS:
Procedure: Indirect Pulp capping-Resin-modified calcium silicate - TheraCal — Use of a dental restorative protocol using Resin-modified calcium silicate - TheraCal pulp capping restorative material
  Arms: Indirect pulp capping therapy-Resin-modified calcium silicate - TheraCal
Procedure: Indirect Pulp capping-Calcium hydroxide - Dycal — Use of a dental restorative protocol using Calcium hydroxide - Dycal pulp capping restorative material
  Arms: Indirect pulp capping therapy- - Calcium hydroxide - Dycal
Procedure: Indirect Pulp capping-Resin-based dentin bonding agent — Use of a dental restorative protocol using resin-based dentin bonding system only
  Arms: Indirect pulp capping therapy-- Resin-based dentin bonding agent
Procedure: Direct Pulp capping-Resin-modified calcium silicate - TheraCal — Use of a dental restorative protocol using Resin-modified calcium silicate - TheraCal pulp capping restorative material
  Arms: Direct pulp capping therapy-Resin-modified calcium silicate - TheraCal
Procedure: Direct Pulp capping-Calcium hydroxide - Dycal — \Use of a dental restorative protocol using Calcium hydroxide - Dycal pulp capping restorative material
  Arms: Direct pulp capping therapy-Resin-modified calcium silicate - Calcium hydroxide - Dycal

SUMMARY:
At present, dentistry aims for conservative treatments with the goal of maintaining as much tooth structure as possible. Dental caries remains the most prevalent chronic disease worldwide; these lesions can progress rapidly and reach deeper areas of the tooth. The carious lesion is considered deep when it goes through the main tissues of the tooth, and it can affect the pulp tissue, where the nerve and nutrients of the tooth are located. There are many treatment options for deep carious lesions and they vary by the clinical scenario. Vital pulp therapy has become a fairly predictable alternative treatment to pulpectomy (root canal therapy). The goal of vital pulp capping therapies is to keep the pulp of the teeth vital to prevent further interventions such as root canal treatments and complex restorative work. There are two main clinical scenarios when treating these lesions, depending on the remaining dentin thickness between the carious lesion and the pulp: vital direct and indirect pulp capping. Direct and indirect vital pulp therapies are routinely performed using different clinical protocols. The clinical protocols are selected based on the remaining dentin (between the tooth preparation and pulp) and the restorative materials. There are few studies that evaluate pulp capping method in adult teeth (permanent dentition); many studies have investigated baby teeth (deciduous teeth). Routine therapies include the using of adhesive restorations with and without an intermediate layer of restorative material. Calcium hydroxide based cements have been used for pulp capping as an intermediate layer of restorative material. More recently a new intermediate layer of restorative material composed of resin-modified calcium silicate has been indicated for use on direct and indirect pulp capping. The aims of this study are to compare, over a period of 12 months, the post-operative sensitivity and pulp vitality of three indirect pulp capping protocols and two direct pulp capping protocol in vital teeth. This study will provide the necessary evidence to allow clinicians to select the best restorative protocol when treating deep carious lesions where indirect and direct pulp capping protocol are needed.

DETAILED DESCRIPTION:
This randomized, controlled, double-blind, prospective study compares over a period of 12 months, the post-operative sensitivity and pulp vitality of three indirect pulp capping protocols (TheraCal, Bisco; Dycal, Caulk, and no liner). The study was approved by the University of Illinois internal review board (Protocol # 2014-1163). Potential subjects will be screened by one of 3 calibrated investigators through a brief interview and intraoral examination. The screening process includes a medical and dental history, demographics, current/concomitant medication, oral soft and hard tissue examination, 2 radiographs: one periapical and one bitewing, and a review of all inclusion and exclusion criteria. The inclusion criteria consist of adults in good general health between 18 and 64 years of age; with primary active carious lesions deep into the dentin (75% or more of carious dentin) of permanent teeth; absence of clinical symptoms of irreversible pulpitis (spontaneous pain and lingering pain for more than 10 seconds after cold stimulus), and absence of periapical pathology, sinus tract, swelling or abnormal mobility. The outcomes measures are pain using visual analog pain scale (pain assessment form) and success rate (pulp vitality based on percussion, palpation, cold test, radiographic findings), collected at the screening visit, intervention day, 24 hours, 7 days, 3 months, 6 months, and 12 months follow-up visits,

ELIGIBILITY:
Inclusion Criteria:

Clinical inclusion criteria:

* Adults in good general health between 18 and 64 years of age;
* Active carious lesions deep into dentin (75% or more of dentin) involving occlusal/incisal and/or proximal surfaces of permanent teeth;
* Absence of clinical symptoms of irreversible pulpitis (spontaneous pain);
* Absence of periapical pathology, sinus tract, swelling or abnormal mobility;
* Restorable teeth.

Radiographic inclusion criteria:

* Extension of carious lesion close to potential exposure upon excavation (within the D3 region - lesion extending 2/3 within dentin); with the presence of a well-defined radiodense zone between the lesion and the pulp;
* Absence of periapical radiolucency;
* Absence of thickening of the periodontal ligament,
* Absence of resorptive defects.

Exclusion Criteria:

* Non restorable teeth;
* Teeth with:
* Recent trauma (within 6 months);
* Calcified root canals;
* Periapical radiolucency;
* Patients experiencing spontaneous moderate to severe pain;
* Patients that are pregnant or planning to become pregnant in the next year.
* Patients taking analgesics, anti-inflammatory, or antidepressant medications;
* Patients with orthodontic treatment;
* Newly erupted teeth.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago College of Dentistry, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was designed to include teeth as participants. If an individual had multiple teeth that met the inclusion criteria, separate consents were signed and teeth were Enrolled. Recruitment was done at the University of Illinois College of Dentistry Comprehensive Adult clinics.
Units Other Than Participants: teeth
Groups:
- Indirect Pulp Capping Therapy-Theracal LC: Group A: Resin-modified calcium silicate - TheraCal LC (Bisco)
- Indirect Pulp Capping Therapy: Calcium Hydroxide - Dycal: Indirect pulp capping therapy-Group B-Calcium hydroxide - Dycal (Dentsply)
- Indirect Pulp Capping-Resin-based Dentin Bonding Agent: Group C: Resin-based dentin bonding agent (All Bond Universal system)
- Direct Pulp Capping Therapy-Theracal LC: Group A: Resin-modified calcium silicate..
- Direct Pulp Capping Therapy: Calcium Hydroxide-Dycal: Direct pulp capping therapy: Calcium hydroxide - Dycal
Period: Overall Study
Arm/Group | Indirect Pulp Capping Therapy-Theracal LC | Indirect Pulp Capping Therapy: Calcium Hydroxide - Dycal | Indirect Pulp Capping-Resin-based Dentin Bonding Agent | Direct Pulp Capping Therapy-Theracal LC | Direct Pulp Capping Therapy: Calcium Hydroxide-Dycal
Started | 25; 30 teeth | 27; 30 teeth | 27; 30 teeth | 10; 10 teeth | 9; 9 teeth
Completed | 21; 25 teeth | 24; 27 teeth | 24; 27 teeth | 6; 6 teeth | 8; 8 teeth
Not Completed | 4; 5 teeth | 3; 3 teeth | 3; 3 teeth | 4; 4 teeth | 1; 1 teeth
Not completed — Lost to Follow-up | 4 | 3 | 3 | 4 | 1

BASELINE CHARACTERISTICS:
Population: The study was designed to include teeth as participants, Baseline Characteristics collected at the unit level.
Units Other Than Participants: Teeth
Groups:
- Indirect Pulp Capping Therapy-Resin-modified Calcium Silicate - TheraCal: Indirect pulp capping therapy-Resin-modified calcium silicate liner - TheraCal (Bisco)
- Indirect Pulp Capping Therapy-Calcium Hydroxide - Dycal: Indirect pulp capping therapy- Calcium hydroxide - Dycal (Dentsply)
- Indirect Pulp Capping Therapy-Resin-based Dentin Bonding Agent: Indirect pulp capping therapy-Resin-based dentin bonding agent (All Bond)
- Direct Pulp Capping Therapy-Resin-modified Calcium Silicate - TheraCal: Direct pulp capping therapy- Resin-modified calcium silicate liner - TheraCal (Bisco)
- Direct Pulp Capping Therapy-Calcium Hydroxide - Dycal: Direct pulp capping therapy: Calcium hydroxide - Dycal (Dentsply)
- Total: Total of all reporting groups
Arm/Group | Indirect Pulp Capping Therapy-Resin-modified Calcium Silicate - TheraCal | Indirect Pulp Capping Therapy-Calcium Hydroxide - Dycal | Indirect Pulp Capping Therapy-Resin-based Dentin Bonding Agent | Direct Pulp Capping Therapy-Resin-modified Calcium Silicate - TheraCal | Direct Pulp Capping Therapy-Calcium Hydroxide - Dycal | Total
Number analyzed (Participants) | 25 | 27 | 27 | 10 | 9 | 98
Number analyzed (Teeth) | 30 | 30 | 30 | 10 | 9 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 27 | 27 | 10 | 9 | 98
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 33.4 [19 to 63] | 39.2 [19 to 63] | 35 [19 to 63] | 39.8 [19 to 63] | 34.9 [19 to 63] | 36.6 [19 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 17 | 4 | 5 | 59
  Male | 9 | 10 | 10 | 6 | 4 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 10 | 8 | 1 | 2 | 24
  Not Hispanic or Latino | 20 | 12 | 15 | 9 | 7 | 63
  Unknown or Not Reported | 2 | 5 | 4 | 0 | 0 | 11
Pulp Diagnosis [Number; unit: Teeth] — Population: Clinical outcome criteria: Pulpal diagnosis: Vital pulp/Nonvital. Vital: (1) palpation ="negative" response. (2) percussion = "negative" response. (3) response to cold stimuli= positive [response time (seconds).
  Non vital: (1) palpation ="positive" response. (2) percussion = "positive"" response. (3) response to cold stimuli= positive or delayed [response time (seconds) and lingering (seconds).
  Teeth
    Vital | 30 | 30 | 30 | 10 | 9 | 109
    Non vital | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Success Rate Based on Pulp Vitality Tests (Vital/Non Vital)
Description: The success rate was based on 3 measures of pulp vitality that resulted in a diagnosis of vital or nonvital after 12-month follow-up:
  Vital: (1) palpation ="negative" response. (2) percussion = "negative" response. (3) response to cold stimuli= positive [response time (seconds).
  Non vital: (1) palpation ="positive" response. (2) percussion = "positive"" response. (3) response to cold stimuli= positive or delayed [response time (seconds) and lingering (seconds).
Time Frame: 12 months
Measure: Number; unit: Percentage of success rate
Units Other Than Participants: Teeth
Groups:
- Indirect Pulp Capping Therapy-Theracal Group; Direct Pulp Capping- Theracal Group: Application of resin-modified calcium silicate (TheraCal LC - Bisco) pulp capping material
- Indirect Pulp Capping Therapy-Dycal Group; Direct Pulp Capping-Dycal Group: Application of calcium hydroxide cement (Dycal - Dentsply) pulp capping material
- Indirect Pulp Capping- No Liner Group: Use of dentin bonding system only. All Bond Universal self-etching system (Bisco)
Arm/Group | Indirect Pulp Capping Therapy-Theracal Group | Indirect Pulp Capping Therapy-Dycal Group | Indirect Pulp Capping- No Liner Group | Direct Pulp Capping- Theracal Group | Direct Pulp Capping-Dycal Group
Number analyzed (Participants) | 21 | 24 | 24 | 6 | 8
Number analyzed (Teeth) | 25 | 27 | 27 | 6 | 8
Percentage of success rate | 96.2 | 100 | 100 | 86 | 100
Statistical Analysis 1: Comparison: Indirect Pulp Capping Therapy-Theracal Group vs Indirect Pulp Capping Therapy-Dycal Group vs Indirect Pulp Capping- No Liner Group vs Direct Pulp Capping- Theracal Group vs Direct Pulp Capping-Dycal Group; The clinical outcome measures assessed were pain using visual analog pain scale, pulp vitality assessment at 12 months. The success rate was based on 3 measures of pulp vitality that resulted in a diagnosis of vital or nonvital: Vital: palpation = negative/ percussion = negative/ response to cold stimuli= positive response Non vital: palpation = positive / percussion = positive. / response to cold stimuli= positive or delayed response time in seconds and lingering; Test type: Superiority — Descriptive data and rates of success were calculated independently for indirect and direct therapies. Statistical analyses of proportions were done using Fisher's test and 95% confidence intervals (CI); p > 0.1, Fisher Exact

2. Primary Outcome: Pain Assessment Using Visual Analog Pain Scale (VAS) Scale.
Description: All the subjects will be asked to answer one question tracing a line on a hard copy visual analogue scale within a centimeters scale (0-10 cm) The measurement was quantitative (cm). The subject is asked to rate the level of pain by drawing a line in a 10 cm line, 0 being no pain, 10 being the worst pain.
Time Frame: 12 months
Measure: Mean (Full Range); unit: cm
Units Other Than Participants: Teeth
Groups:
- Indirect Pulp Capping Therapy-Theracal Group: Application of resin-modified calcium silicate (TheraCal - Bisco) pulp capping material
- Indirect Pulp Capping Therapy- Dycal Group: Application of Calcium hydroxide pulp capping cement (Dycal - Dentsply) pulp capping material
- Indirect Pulp Capping- Dentin Bonding Agent: Use of dentin bonding system All Bond Universal self-etching system (Bisco)
- Direct Pulp Capping- Theracal Group: Application of resin modified calcium silicate (Theracal - Bisco) pulp capping material
- Direct Pulp Capping- Dycal Group: Application of calcium hydroxide cement (Dycal - Dentsply) pulp capping material
Arm/Group | Indirect Pulp Capping Therapy-Theracal Group | Indirect Pulp Capping Therapy- Dycal Group | Indirect Pulp Capping- Dentin Bonding Agent | Direct Pulp Capping- Theracal Group | Direct Pulp Capping- Dycal Group
Number analyzed (Participants) | 21 | 24 | 24 | 6 | 8
Number analyzed (Teeth) | 25 | 27 | 27 | 6 | 8
cm | 0 [0 to 0] | 0.7 [0 to 2] | 1.6 [0 to 4.1] | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Indirect Pulp Capping -Resin-modified Calcium Silicate - TheraCal LC: Indirect pulp capping - Resin-modified calcium silicate liner - TheraCal LC
- Indirect Pulp Capping -Calcium Hydroxide - Dycal: Indirect pulp capping - Calcium hydroxide - Dycal
- Indirect Pulp Capping- Resin-based Dentin Bonding Agent: Indirect pulp capping Resin-based dentin bonding agent- (All bond)
- Direct Pulp Capping -Resin-modified Calcium Silicate - TheraCal LC: Direct pulp capping Resin-modified calcium silicate - TheraCal LC
- Direct Pulp Capping-Calcium Hydroxide - Dycal: Direct pulp capping Calcium hydroxide - Dycal
Arm/Group | Indirect Pulp Capping -Resin-modified Calcium Silicate - TheraCal LC | Indirect Pulp Capping -Calcium Hydroxide - Dycal | Indirect Pulp Capping- Resin-based Dentin Bonding Agent | Direct Pulp Capping -Resin-modified Calcium Silicate - TheraCal LC | Direct Pulp Capping-Calcium Hydroxide - Dycal
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/10 | 0/9

LIMITATIONS AND CAVEATS:
Not all participants completed 100% of the follow-ups. Limited numbers of participants in the direct pulp capping study arm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT02635867/Prot_SAP_000.pdf